CLINICAL TRIAL: NCT02996500
Title: A 12 WEEK RANDOMIZED, DOUBLE-BLIND, DOUBLE DUMMY, PARALLEL GROUP, ACTIVE AND PLACEBO-CONTROLLED, MULTICENTER STUDY TO ASSESS THE EFFICACY AND SAFETY PROFILE OF PF-06650833 IN SUBJECTS WITH ACTIVE RHEUMATOID ARTHRITIS WITH AN INADEQUATE RESPONSE TO METHOTREXATE
Brief Title: Safety and Efficacy of Pf-06650833 In Subjects With Rheumatoid Arthritis, With An Inadequate Response To Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B7921005; 2016-002337-30 (EudraCT Number); IRAK 4 (Other: Alias Study Number)
Record Dates: First submitted 2016-10-13; First posted 2016-12-19 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide; tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1: 20 mg QD (Experimental): PF-06650833 , 20 mg QD
  Interventions: Drug: PF-06650833
- Arm 2: 60 mg QD (Experimental): PF-06650833, 60 mg QD
  Interventions: Drug: PF-06650833
- Arm 3: 200 mg QD (Experimental): Pf-06650833, 200 mg QD
  Interventions: Drug: PF-06650833
- Arm 4: 400 mg QD (Experimental): PF-06650833, 400 mg QD
  Interventions: Drug: PF-06650833
- Placebo (Placebo Comparator): Placebo, 0 mg BID
  Interventions: Drug: Placebo
- Arm 5: Tofacitinib (Active Comparator): Tofacitinib 5 mg BID
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: PF-06650833 — Investigational
  Arms: Arm 1: 20 mg QD; Arm 2: 60 mg QD; Arm 3: 200 mg QD; Arm 4: 400 mg QD
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Tofacitinib — Investigational
  Other Names: Xeljanz
  Arms: Arm 5: Tofacitinib

SUMMARY:
This is a Phase 2, multicenter, randomized, double blind, double dummy, placebo and active-controlled, parallel group study to assess the efficacy and safety of PF 06650833 at Week 12 in subjects with moderate-severe, active, RA who have had an inadequate response to MTX. PF-06650833 or matching placebo tablets will be administered orally QD under fasting conditions, and tofacitinib or matching tofacitinib placebo tablets will be administered orally BID for 12 weeks in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female (including WOCBP) subjects between the ages of 18 and 75 years, inclusive.
2. Diagnosis of RA and meeting the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for RA with a Total Score ≥6/10.
3. The subject has active disease at both Screening and Baseline, as defined by both:

   * 6 joints tender or painful on motion, AND
   * 6 joints swollen; and fulfills 1 of the following 2 criteria at Screening:
   * High sensitivity C reactive protein (hsCRP) >7 mg/L at screening
   * Erythrocyte sedimentation rate (ESR) (Westergren method) >28 mm/hr;
4. Meets Class I, II or III of the ACR 1991 Revised Criteria for Global Functional Status in RA.
5. Subjects must be ACPA positive between screening and randomization.
6. Subjects must have been taking oral MTX for at least 3 months at an adequate dose to determine that the subject had an inadequate response to MTX
7. Up to 50 % of subjects may have received one (and only one) approved TNF-inhibiting biologic agent administered that was inadequately effective and/or not tolerated. The anti-TNF biologic could also have been discontinued due to lack of continued access.

Exclusion Criteria:

1. Subjects with a known immunodeficiency disorder or a first degree relative with a hereditary immunodeficiency.
2. Subjects with any of the following infections or infections history:

   1. Any infection requiring treatment within 2 weeks prior to screening (Visit 1).
   2. Any infection requiring hospitalization, parenteral antimicrobial therapy within 60 days, or as otherwise judged to be an opportunistic infection or clinically significant by the investigator, within the past 6 months.
   3. Infected joint prosthesis at any time with the prosthesis still in situ.
   4. Recurrent (more than one episode) herpes zoster or disseminated (a single episode) herpes zoster or disseminated (a single episode) herpes simplex.
   5. Subjects will be screened for HIV. Subjects who test positive for HIV will be excluded from the study.
   6. Subjects will be screened for hepatitis B virus infection and will be excluded if positive for hepatitis B surface antigen (HBsAg). Subjects with HBsAg negative testing but who test positive for hepatitis B core antibody (HBcAb) must have further testing for hepatitis B surface antibody (HBsAb). If HBsAb is negative, the subject will be excluded from the study.
   7. Subjects with clinically significant active hepatic disease or hepatic impairment by laboratory assessment.
   8. Subjects will be screened for hepatitis C virus (HCV Ab). Subjects with positive HCV Ab tests will be reflex tested for HCV ribonucleic acid (HCV RNA). Only subjects with negative HCV Ab or HCV RNA will be allowed to enroll in the study.
3. Evidence of active or latent, untreated or inadequately treated infection with Mycobacterium tuberculosis (TB)
4. Pre-existing chronic autoimmune disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (100):
- United States (14):
  - Clinical and Translational Research Center of Alabama, PC, Tuscaloosa, Alabama
  - Dory Hardy, PharmD, Tucson, Arizona
  - Southern Arizona VA Health care System, Tucson, Arizona
  - Robert W. Levin, MD,PA, Clearwater, Florida
  - Millennium Research, Ormond Beach, Florida
  - Arthritis & Rheumatic Care Center, South Miami, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - Medical Associates of North Georgia, Canton, Georgia
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Arthritis and Diabetes Clinic, Inc., Monroe, Louisiana
  - Ramesh C Gupta, M.D., Memphis, Tennessee
  - Accurate Clinical Management, LLC, Baytown, Texas
  - Accurate Clinical Management, LLC, Houston, Texas
  - DM Clinical Research, Tomball, Texas
- Australia (2):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Genesis Research Services, Broadmeadow, New South Wales
- Bosnia and Herzegovina (3):
  - General Hospital "Prim.dr.Abdulah Nakas", Sarajevo, Kanton Sarajevo
  - University Clinical Center Republic of Srpska, Banja Luka, Republika Srpska
  - Health Center Gradiska, Gradiška, Republika Srpska
- Bulgaria (5):
  - UMHAT Kaspela, Plovdiv
  - MHAT Liulin, Sofia
  - UMHAT "Sv.Ivan Rilski", Clinic of rheumatology, Sofia
  - Medical Center Synexus Sofia EOOD, Sofia
  - Specialized Hospital for Active Treatment of Oncology Diseases EAD, Department of Imaging Diagnostic, Sofia
- Croatia (2):
  - Poliklinika K-centar, Zagreb, City of Zagreb
  - Medicinski centar Kuna&Peric, Zagreb
- Czechia (3):
  - CCBR Ostrava s.r.o., Ostrava
  - Revmatologicka ambulance, Prague
  - Medical Plus s.r.o., Uherské Hradiště
- Georgia (7):
  - LTD Israeli-Georgian Medical Research Clinic HELSICORE, Tbilisi
  - LTD " Diagnostic Service ", Tbilisi
  - Ltd Institute of Clinical Cardiology, Tbilisi
  - LTD Unimedi Kakheti, Tbilisi
  - LTD "MediClubGeorgia", Tbilisi
  - Ltd "Medicore", Tbilisi
  - Unimedi Kakheti LTD, Telavi
- Knappschaftsklinikum Saar GmbH, Püttlingen, Germany
- Hungary (6):
  - Revita Reumatologiai Rendelo, Budapest
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - CRU Hungary Ltd., Miskolc
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Mozgasszervi Rehabilitacios Osztaly, Szentes
  - VITAL MEDICAL CENTER Orvosi es Fogorvosi Kozpont, Veszprém
- Mexico (4):
  - Private Practice - Dr. Miguel Cortes Hernandez, Cuernavaca, Morelos
  - Centro Peninsular de Investigacion Clinica S.C.P, Mérida, Yucatán
  - Kohler & Milstein Research S.A de C.V, Mérida, Yucatán
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosi, S.C., San Luis Potosí City
- Poland (9):
  - Szpital Specjalistyczny nr 1 w Bytomiu, Bytom
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Synexus Polska Sp z o.o. Oddzial w Gdyni, Gdynia
  - McBk S.C., Grodzisk Mazowiecki
  - Synexus Polska Sp.Zo.o., Katowice
  - Prywatna Praktyka Lekarska Prof. UM Dr hab. Med. Pawel Hrycaj, Poznan
  - Synexus Polska Sp. z o.o., Warsaw
  - Reumatika Centrum Reumatologii NZOZ, Warsaw
  - Synexus Polska Sp. z o.o. Oddział we Wroclawiu, Wroclaw
- Romania (6):
  - Centrul Medical Unirea, Bucharest
  - Med Life, Bucharest
  - Centrul Medical Sana, Bucharest
  - Euroclinic Hospital, Bucharest
  - Spitalul Clinic de Recuperare Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Tirgu Mures, Târgu Mureş
- Russia (8):
  - FSBEI HE "Kazan State Medical University" MoH of RF, Kazan'
  - FSBSI "Scientific Research Institute of Rheumatology n.a. V.A. Nasonova", Moscow
  - SBHI of Moscow City Clinical Hospital # 1 n.a. N.I. Pirogov of Moscow Healthcare Department, Moscow
  - FSBHI Central Clinical Hospital of Russian Academy of Sciences, Moscow
  - State Budgetary Institution of Ryazan Region "Regional clinical cardiology dispensary", Ryazan
  - LLC "Sanavita", Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Health Care "Clinical Rheumatology Hospital #25", Saint Petersburg
  - SBHI of VR "Regional Clinical Hospital", Vladimir
- Serbia (4):
  - Institute of Rheumatology, Belgrade
  - Military Medical Academy, Belgrade
  - Institute for Treatment and Rehabilitation "Niska Banja", Niška Banja
  - Special Hospital for Rheumatic Diseases Novi Sad, Novi Sad
- Slovakia (6):
  - Reumacentrum s.r.o., Partizánske, Trenčín Region
  - AAGS s.r.o., Reumatologicka ambulancia, Dunajská Streda
  - Nemocnica Kosice-Saca, a.s.1.sukromna nemocnica, Kosice-Saca
  - Neštátna Reumatologická ambulancia, Považská Bystrica
  - REUMEX s.r.o. Reumatologicka ambulancia, Rimavská Sobota
  - Reumatologicka ambulancia, MUDr. Pavol Polak s.r.o., Žilina
- South Korea (4):
  - Seoul National University hospital, Seoul
  - Hanyang University Seoul hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
- Spain (5):
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - HM Hospital Nuestra Señora de La Esperanza, Santiago de Compostela, A Coruña
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Quironsalud Infanta Luisa, Seville
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
- Ukraine (8):
  - Komunalnyi likuvalno-profilaktychnyi zaklad "Chernihivska oblasna likarnia",, Chernihiv
  - Derzhavna ustanova "Natsionalnyi instytut terapii imeni L.T. Maloi, Kharkiv
  - Komunalne nekomertsiine pidpryiemstvo "Konsultatyvno-diahnostychnyi tsentr", Kyiv
  - Medychnyi tsentr tovarystva z obmezhenoiu vidpovidalnistiu "Revmotsentr", m. Kyiv, Kyiv
  - Derzhavna ustanova "Instytut herontolohii imeni D.F. Chebotarova, Kyiv
  - Poltavska oblasna klinichna likarnia im. M.V. Sklifosovskoho,, Poltava
  - Ternopilska universytetska likarnia, revmatolohichne viddilennia, Derzhavnyi vyshchyi navchalnyi, Ternopil
  - Vinnytska oblasna klinichna likarnia im. M.I.Pyrohova, revmatolohichne viddilennia, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7921005

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received 4 matching PF-06650833 modified release (MR) placebo tablets once daily (QD) and 1 matching tofacitinib placebo tablet twice a day (BID) in 12 weeks treatment period.
- Tofa 10 mg: Participants received 4 matching PF-06650833 MR placebo tablets QD and tofacitinib (Tofa) 10 mg (5 mg tablet BID) in 12 weeks treatment period.
- PF-06650833 20 mg: Participants received 1 MR tablet of PF-06650833 20 mg and 3 matching PF-06650833 MR placebo tablets QD, 1 matching tofacitinib placebo tablet BID in 12 weeks treatment period.
- PF-06650833 60 mg: Participants received 3 MR tablets of PF-06650833 20 mg and 1 matching PF-06650833 MR placebo tablet QD, 1 matching tofacitinib placebo tablet BID in 12 weeks treatment period.
- PF-06650833 200 mg: Participants received 2 MR tablets of PF-06650833 100 mg and 2 matching PF-06650833 MR placebo tablets QD, 1 matching tofacitinib placebo tablet BID in 12 weeks treatment period.
- PF-06650833 400 mg: Participants received 4 MR tablets of PF-06650833 100 mg QD and 1 matching tofacitinib placebo tablet BID in 12 weeks treatment period.
Period: Overall Study
Arm/Group | Placebo | Tofa 10 mg | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Started | 39 | 43 | 39 | 50 | 50 | 48
Completed | 31 | 42 | 29 | 46 | 45 | 44
Not Completed | 8 | 1 | 10 | 4 | 5 | 4
Not completed — Adverse Event | 1 | 1 | 4 | 3 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 1
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Non-Compliance With Study Drug | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 3 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population was defined as all participants who were randomized to study treatment and received at least 1 dose of the randomized investigational drug (PF-06650833, tofacitinib, or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tofa 10 mg | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg | Total
Number analyzed (Participants) | 39 | 43 | 39 | 50 | 50 | 48 | 269
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (10.51) | 52.7 (10.02) | 55.9 (9.74) | 51.0 (12.05) | 53.6 (11.47) | 54.8 (8.76) | 53.7 (10.56)
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 7 | 9 | 5 | 15 | 11 | 6 | 53
  45-64 Years | 26 | 29 | 27 | 29 | 32 | 36 | 179
  >=65 Years | 6 | 5 | 7 | 6 | 7 | 6 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 31 | 42 | 39 | 37 | 210
  Male | 9 | 12 | 8 | 8 | 11 | 11 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 37 | 43 | 37 | 47 | 47 | 43 | 254
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 1 | 2 | 2 | 8
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 1 | 1 | 0 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Simplified Disease Activity Index (SDAI) at Week 12
Description: The SDAI is a continuous composite measure derived from components of the American College of Rheumatology (ACR) Core Dataset.The SDAI was calculated using the following formula: SDAI = Tender / Painful Joint Count(TJC) (using 28 joints) + Swollen Joint Count (SJC) (using 28 joints) + Patient Global Assessment of Arthritis (PtGA) (0-10 cm scale) + Physician's Global Assessment of Arthritis (PhGA) (0-10 cm scale) + high sensitivity C-reactive protein (hsCRP) (mg/dL). SDAI total score= 0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity. The primary analysis utilized a Bayesian ANCOVA model with an informative placebo prior distribution with borrowing from tofacitinib historical placebo data. The confidence interval was credible interval in this statistical analysis. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline and Week 12
Population: The analysis population included all participants who were randomized to the study, received at least 1 dose of the randomized investigational drug (PF-06650833, or placebo), and had data collected for this outcome measure at the time points assessed. It was pre-specified in the protocol to not summarize this efficacy endpoint for Tofa arm.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- PF-06650833 400 mg: Participants received 4 modified release (MR) tablets of PF-06650833 400 mg once daily (QD) and 1 matching tofacitinib placebo tablet twice a day (BID) in 12 weeks treatment period.
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 34 | 30 | 45 | 44 | 45
units on a scale | -13.87 [-17.70 to -10.02] | -21.71 [-26.14 to -17.20] | -22.83 [-26.57 to -19.20] | -24.77 [-28.54 to -21.08] | -25.16 [-28.85 to -21.39]
Statistical Analysis 1: Comparison: Placebo vs PF-06650833 20 mg; The confidence interval was credible interval in this analysis; Test type: Superiority; p = 0.0050, ANCOVA; Bayesian analysis of covariance (ANCOVA) modeling framework was used with baseline SDAI score as a covariate; Mean Difference (Net) = -7.83, 95% CI 2-sided [-13.73 to -1.97]
Statistical Analysis 2: Comparison: Placebo vs PF-06650833 60 mg; The confidence interval was credible interval in this analysis; Test type: Superiority; p < 0.001, ANCOVA; Bayesian analysis of covariance (ANCOVA) modeling framework was used with baseline SDAI score as a covariate; Mean Difference (Net) = -8.96, 95% CI 2-sided [-14.37 to -3.66]
Statistical Analysis 3: Comparison: Placebo vs PF-06650833 200 mg; The confidence interval was credible interval in this analysis; Test type: Superiority; p < 0.001, ANCOVA; Bayesian analysis of covariance (ANCOVA) modeling framework was used with baseline SDAI score as a covariate; Median Difference (Net) = -10.89, 95% CI 2-sided [-16.36 to -5.63]
Statistical Analysis 4: Comparison: Placebo vs PF-06650833 400 mg; The confidence interval was credible interval in this analysis; Test type: Superiority; p < 0.001, ANCOVA; Bayesian analysis of covariance (ANCOVA) modeling framework was used with baseline SDAI score as a covariate; Mean Difference (Net) = -11.29, 95% CI 2-sided [-16.62 to -5.92]

2. Secondary Outcome: Change From Baseline in SDAI at Weeks 4 and 8
Description: The SDAI is a continuous composite measure derived from components of the American College of Rheumatology (ACR) Core Dataset.The SDAI was calculated using the following formula: SDAI = TJC (using 28 joints) + SJC (using 28 joints) + PtGA (0-10 cm scale) + PhGA (0-10 cm scale) + hsCRP (mg/dL). SDAI total score= 0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity. The descriptive summary of change from baseline in SDAI was based on a mixed effect model repeat measurement MMRM model with observed data. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4 and 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  Week 4: number analyzed (Participants) | 37 | 37 | 49 | 47 | 47
  Week 4 | -10.78 [-15.07 to -6.49] | -12.39 [-14.68 to -10.10] | -14.29 [-16.87 to -11.71] | -13.56 [-17.25 to -9.86] | -12.30 [-15.46 to -9.14]
  Week 8: number analyzed (Participants) | 34 | 34 | 46 | 41 | 45
  Week 8 | -17.07 [-22.58 to -11.55] | -16.62 [-20.71 to -12.53] | -18.85 [-22.03 to -15.67] | -19.95 [-24.81 to -15.08] | -21.15 [-25.50 to -16.79]

3. Secondary Outcome: Percentage of Participants With SDAI Low Disease Activity Score (LDAS) (SDAI <=11) at 4, 8, and 12 Weeks
Description: The SDAI is a continuous composite measure derived from components of the American College of Rheumatology (ACR) Core Dataset.The SDAI was calculated using the following formula: SDAI = TJC (using 28 joints) + SJC (using 28 joints) + PtGA (0-10 cm scale) + PhGA (0-10 cm scale) + hsCRP (mg/dL). The criterion of SDAI LDAS was SDAI<=11. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 47 | 47
  Week 4 | 8.1 [0.0 to 16.9] | 7.9 [0.0 to 16.5] | 12.2 [3.1 to 21.4] | 10.6 [1.8 to 19.5] | 8.5 [0.5 to 16.5]
  Week 8: number analyzed (Participants) | 34 | 35 | 46 | 41 | 45
  Week 8 | 14.7 [2.8 to 26.6] | 20.0 [6.7 to 33.3] | 17.4 [6.4 to 28.3] | 29.3 [15.3 to 43.2] | 33.3 [19.6 to 47.1]
  Week 12: number analyzed (Participants) | 34 | 31 | 45 | 44 | 45
  Week 12 | 26.5 [11.6 to 41.3] | 41.9 [24.6 to 59.3] | 28.9 [15.6 to 42.1] | 38.6 [24.2 to 53.0] | 42.2 [27.8 to 56.7]

4. Secondary Outcome: Percentage of Participants With SDAI Remission (SDAI <=3.3) at 4, 8, and 12 Weeks
Description: The SDAI is a continuous composite measure derived from components of the American College of Rheumatology (ACR) Core Dataset.The SDAI was calculated using the following formula: SDAI = TJC (using 28 joints) + SJC (using 28 joints) + PtGA (0-10 cm scale) + PhGA (0-10 cm scale) + hsCRP (mg/dL). The criterion of SDAI remission was SDAI<=3.3. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 47 | 47
  Week 4 | 0 [0.0 to 0.0] | 2.6 [0.0 to 7.7] | 2.0 [0.0 to 6.0] | 0 [0.0 to 0.0] | 2.1 [0.0 to 6.3]
  Week 8: number analyzed (Participants) | 34 | 35 | 46 | 41 | 45
  Week 8 | 0 [0.0 to 0.0] | 8.6 [0.0 to 17.8] | 0 [0.0 to 0.0] | 7.3 [0.0 to 15.3] | 2.2 [0.0 to 6.5]
  Week 12: number analyzed (Participants) | 34 | 31 | 45 | 44 | 45
  Week 12 | 2.9 [0.0 to 8.6] | 3.2 [0.0 to 9.4] | 2.2 [0.0 to 6.5] | 6.8 [0.0 to 14.3] | 8.9 [0.6 to 17.2]

5. Secondary Outcome: Percentage of Participants With Disease Activity Score-28 (4 Components Based on Erythrocyte Sedimentation Rate) (DAS28-4 [ESR]) LDAS (DAS28 <3.2) at 4, 8, and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-4 (ESR) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed, ESR and PGA. DAS28-4 (ESR) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.70 ln(ESR [mm/first hour] + 0.014 (PtGA [mm]). Total score range: 0-9.4. Higher score indicated more disease activity. The criterion of DAS28-4 (ESR) LDAS was DAS28<3.2. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 35 | 37 | 47 | 48 | 47
  Week 4 | 2.9 [0.0 to 8.4] | 8.1 [0.0 to 16.9] | 6.4 [0.0 to 13.4] | 8.3 [0.5 to 16.2] | 4.3 [0.0 to 10.0]
  Week 8: number analyzed (Participants) | 35 | 35 | 44 | 45 | 47
  Week 8 | 8.6 [0.0 to 17.8] | 17.1 [4.7 to 29.6] | 13.6 [3.5 to 23.8] | 13.3 [3.4 to 23.3] | 12.8 [3.2 to 22.3]
  Week 12: number analyzed (Participants) | 34 | 30 | 45 | 45 | 45
  Week 12 | 17.6 [4.8 to 30.5] | 20.0 [5.7 to 34.3] | 24.4 [11.9 to 37.0] | 22.2 [10.1 to 34.4] | 17.8 [6.6 to 28.9]

6. Secondary Outcome: Percentage of Participants With DAS28-3 (ESR) LDAS (DAS28 <3.2) at 4, 8, and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-3 (ESR) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed and ESR. DAS28-3 (ESR) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.70 ln(ESR [mm/first hour]*1.08+0.16. Total score range: 0-9.4. Higher score indicated more disease activity. The criterion of DAS28-3 LDAS was DAS28<3.2. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 35 | 37 | 47 | 48 | 47
  Week 4 | 5.7 [0.0 to 13.4] | 8.1 [0.0 to 16.9] | 10.6 [1.8 to 19.5] | 8.3 [0.5 to 16.2] | 4.3 [0.0 to 10.0]
  Week 8: number analyzed (Participants) | 35 | 35 | 44 | 45 | 47
  Week 8 | 8.6 [0.0 to 17.8] | 20.0 [6.7 to 33.3] | 15.9 [5.1 to 26.7] | 8.9 [0.6 to 17.2] | 14.9 [4.7 to 25.1]
  Week 12: number analyzed (Participants) | 34 | 30 | 45 | 45 | 45
  Week 12 | 20.6 [7.0 to 34.2] | 20.0 [5.7 to 34.3] | 22.2 [10.1 to 34.4] | 22.2 [10.1 to 34.4] | 15.6 [5.0 to 26.1]

7. Secondary Outcome: Percentage of Participants With Disease Activity Score-28 (4 Components Based on High-Sensitivity C-Reactive Protein) (DAS28-4 [CRP]) LDAS (DAS28 <3.2) at 4, 8, and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-4 (CRP) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed, hs-CRP and PtGA. DAS28-4 (CRP) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 ln(CRP [mg/L] +1) + 0.014 (PtGA [mm]) + 0.96. Total score range: 0-9.4. Higher score indicated more disease activity. The criterion of DAS28-4 LDAS was DAS28<3.2. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 47 | 47
  Week 4 | 8.1 [0.0 to 16.9] | 13.2 [2.4 to 23.9] | 16.3 [6.0 to 26.7] | 12.8 [3.2 to 22.3] | 8.5 [0.5 to 16.5]
  Week 8: number analyzed (Participants) | 34 | 35 | 46 | 41 | 45
  Week 8 | 11.8 [0.9 to 22.6] | 20.0 [6.7 to 33.3] | 19.6 [8.1 to 31.0] | 26.8 [13.3 to 40.4] | 33.3 [19.6 to 47.1]
  Week 12: number analyzed (Participants) | 34 | 31 | 45 | 44 | 45
  Week 12 | 20.6 [7.0 to 34.2] | 38.7 [21.6 to 55.9] | 35.6 [21.6 to 49.5] | 40.9 [26.4 to 55.4] | 42.2 [27.8 to 56.7]

8. Secondary Outcome: Percentage of Participants With DAS28-3 (CRP) LDAS (DAS28 <3.2) at 4, 8, and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-3 (CRP) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed and hs-CRP. DAS28-3 (CRP) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 ln(CRP [mg/L] +1)*1.10+ 1.15. Total score range: 0-9.4. Higher score indicated more disease activity. The criterion of DAS28-3 LDAS was DAS28<3.2. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 47 | 47
  Week 4 | 8.1 [0.0 to 16.9] | 10.5 [0.8 to 20.3] | 16.3 [6.0 to 26.7] | 17.0 [6.3 to 27.8] | 10.6 [1.8 to 19.5]
  Week 8: number analyzed (Participants) | 34 | 35 | 46 | 41 | 45
  Week 8 | 20.6 [7.0 to 34.2] | 22.9 [8.9 to 36.8] | 19.6 [8.1 to 31.0] | 34.1 [19.6 to 48.7] | 37.8 [23.6 to 51.9]
  Week 12: number analyzed (Participants) | 34 | 31 | 45 | 44 | 45
  Week 12 | 23.5 [9.3 to 37.8] | 41.9 [24.6 to 59.3] | 40.0 [25.7 to 54.3] | 47.7 [33.0 to 62.5] | 42.2 [27.8 to 56.7]

9. Secondary Outcome: Percentage of Participants With DAS28-4 (ESR) Remission (DAS28 <2.6) at 4, 8 and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-4 (ESR) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed, ESR and PtGA. DAS28-4 (ESR) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.70 ln(ESR [mm/first hour] + 0.014 (PtGA [mm]). Total score range: 0-9.4. Higher score indicated more disease activity. The criterion of DAS28-4 remission was DAS28<2.6. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 35 | 37 | 47 | 48 | 47
  Week 4 | 0 [0.0 to 0.0] | 5.4 [0.0 to 12.7] | 2.1 [0.0 to 6.3] | 8.3 [0.5 to 16.2] | 2.1 [0.0 to 6.3]
  Week 8: number analyzed (Participants) | 35 | 35 | 44 | 45 | 47
  Week 8 | 5.7 [0.0 to 13.4] | 11.4 [0.9 to 22.0] | 9.1 [0.6 to 17.6] | 6.7 [0.0 to 14.0] | 10.6 [1.8 to 19.5]
  Week 12: number analyzed (Participants) | 34 | 30 | 45 | 45 | 45
  Week 12 | 5.9 [0.0 to 13.8] | 16.7 [3.3 to 30.0] | 13.3 [3.4 to 23.3] | 8.9 [0.6 to 17.2] | 11.1 [1.9 to 20.3]

10. Secondary Outcome: Percentage of Participants With DAS28-3 (ESR) Remission (DAS28 <2.6) at 4, 8 and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-3 (ESR) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed and ESR. DAS28-3 (ESR) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.70 ln(ESR [mm/first hour]*1.08+0.16. Total score range: 0-9.4. Higher score indicated more disease activity. The criterion of DAS28-3 remission was DAS28<2.6. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 35 | 37 | 47 | 48 | 47
  Week 4 | 0 [0.0 to 0.0] | 2.7 [0.0 to 7.9] | 2.1 [0.0 to 6.3] | 6.3 [0.0 to 13.1] | 2.1 [0.0 to 6.3]
  Week 8: number analyzed (Participants) | 35 | 35 | 44 | 45 | 47
  Week 8 | 2.9 [0.0 to 8.4] | 8.6 [0.0 to 17.8] | 9.1 [0.6 to 17.6] | 6.7 [0.0 to 14.0] | 8.5 [0.5 to 16.5]
  Week 12: number analyzed (Participants) | 34 | 30 | 45 | 45 | 45
  Week 12 | 8.8 [0.0 to 18.4] | 10.0 [0.0 to 20.7] | 13.3 [3.4 to 23.3] | 11.1 [1.9 to 20.3] | 8.9 [0.6 to 17.2]

11. Secondary Outcome: Percentage of Participants With DAS28-4 (CRP) Remission (DAS28 <2.6) at 4, 8 and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-4 (CRP) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed, hs-CRP and PtGA. DAS28-4 (CRP) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 ln(CRP [mg/L] +1) + 0.014 (PtGA [mm]) + 0.96. Total score range: 0-9.4. Higher score indicated more disease activity. The criterion of DAS28-4 remission was DAS28<2.6. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 47 | 47
  Week 4 | 2.7 [0.0 to 7.9] | 5.3 [0.0 to 12.4] | 8.2 [0.5 to 15.8] | 10.6 [1.8 to 19.5] | 6.4 [0.0 to 13.4]
  Week 8: number analyzed (Participants) | 34 | 35 | 46 | 41 | 45
  Week 8 | 8.8 [0.0 to 18.4] | 17.1 [4.7 to 29.6] | 10.9 [1.9 to 19.9] | 22.0 [9.3 to 34.6] | 13.3 [3.4 to 23.3]
  Week 12: number analyzed (Participants) | 34 | 31 | 45 | 44 | 45
  Week 12 | 14.7 [2.8 to 26.6] | 22.6 [7.9 to 37.3] | 17.8 [6.6 to 28.9] | 25.0 [12.2 to 37.8] | 24.4 [11.9 to 37.0]

12. Secondary Outcome: Percentage of Participants With DAS28-3 (CRP) Remission (DAS28 <2.6) at 4, 8 and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-3 (CRP) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed and hs-CRP. DAS28-3 (CRP) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 ln(CRP [mg/L] +1)*1.10+1.15. Total score range: 0-9.4. Higher score indicated more disease activity. The criterion of DAS28-3 remission was DAS28<2.6. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 47 | 47
  Week 4 | 5.4 [0.0 to 12.7] | 5.3 [0.0 to 12.4] | 10.2 [1.7 to 18.7] | 8.5 [0.5 to 16.5] | 4.3 [0.0 to 10.0]
  Week 8: number analyzed (Participants) | 34 | 35 | 46 | 41 | 45
  Week 8 | 8.8 [0.0 to 18.4] | 14.3 [2.7 to 25.9] | 10.9 [1.9 to 19.9] | 22.0 [9.3 to 34.6] | 13.3 [3.4 to 23.3]
  Week 12: number analyzed (Participants) | 34 | 31 | 45 | 44 | 45
  Week 12 | 11.8 [0.9 to 22.6] | 25.8 [10.4 to 41.2] | 22.2 [10.1 to 34.4] | 22.7 [10.3 to 35.1] | 22.2 [10.1 to 34.4]

13. Secondary Outcome: Change From Baseline in DAS28-4 (ESR) at 4, 8 and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-4 (ESR) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed, ESR and PtGA. DAS28-4 (ESR) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.70 ln(ESR [mm/first hour] + 0.014 (PtGA [mm]). Higher score indicated more disease activity. Total score range: 0-9.4. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: The analysis population included all participants who were randomized to the study, received at least 1 dose of the randomized investigational drug (PF-06650833, or placebo), and had data collected for this outcome measure at the time points assessed.It was pre-specified in the protocol to not summarize this efficacy endpoint for Tofa arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  Week 4: number analyzed (Participants) | 35 | 37 | 47 | 48 | 47
  Week 4 | -0.80 [-1.13 to -0.47] | -1.15 [-1.47 to -0.82] | -1.35 [-1.64 to -1.07] | -1.14 [-1.42 to -0.86] | -1.13 [-1.42 to -0.84]
  Week 8: number analyzed (Participants) | 35 | 35 | 44 | 45 | 47
  Week 8 | -1.38 [-1.80 to -0.97] | -1.59 [-2.01 to -1.17] | -1.92 [-2.29 to -1.56] | -1.77 [-2.14 to -1.41] | -2.01 [-2.37 to -1.64]
  Week 12: number analyzed (Participants) | 34 | 30 | 45 | 45 | 45
  Week 12 | -1.55 [-1.97 to -1.13] | -1.85 [-2.28 to -1.41] | -2.37 [-2.74 to -2.01] | -2.23 [-2.60 to -1.86] | -2.36 [-2.73 to -1.99]

14. Secondary Outcome: Change From Baseline in DAS28-3 (ESR) at 4, 8 and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-3 (ESR) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed and ESR. DAS28-3 (ESR) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.70 ln(ESR) [mm/first hour]*1.08+0.16. Total score range: 0-9.4. Higher score indicated more disease activity. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  Week 4: number analyzed (Participants) | 35 | 37 | 47 | 48 | 47
  Week 4 | -0.69 [-1.01 to -0.38] | -1.08 [-1.39 to -0.77] | -1.25 [-1.52 to -0.97] | -1.08 [-1.35 to -0.80] | -1.02 [-1.29 to -0.74]
  Week 8: number analyzed (Participants) | 35 | 35 | 44 | 45 | 47
  Week 8 | -1.14 [-1.54 to -0.75] | -1.52 [-1.92 to -1.12] | -1.80 [-2.15 to -1.45] | -1.62 [-1.97 to -1.27] | -1.79 [-2.14 to -1.44]
  Week 12: number analyzed (Participants) | 34 | 30 | 45 | 45 | 45
  Week 12 | -1.31 [-1.71 to -0.92] | -1.69 [-2.09 to -1.28] | -2.26 [-2.60 to -1.91] | -2.05 [-2.40 to -1.71] | -2.04 [-2.38 to -1.69]

15. Secondary Outcome: Change From Baseline in DAS28-4 (CRP) at 4, 8 and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-4 (CRP) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed, hs-CRP and PtGA. DAS28-4 (CRP) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 ln(CRP [mg/L] +1) + 0.014 (PtGA [mm]) + 0.96. Total score range: 0-9.4. Higher score indicated more disease activity. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 47 | 47
  Week 4 | -0.72 [-1.02 to -0.42] | -0.99 [-1.29 to -0.69] | -1.21 [-1.47 to -0.94] | -1.08 [-1.34 to -0.81] | -0.99 [-1.25 to -0.72]
  Week 8: number analyzed (Participants) | 34 | 35 | 46 | 41 | 45
  Week 8 | -1.20 [-1.58 to -0.83] | -1.31 [-1.68 to -0.94] | -1.59 [-1.92 to -1.27] | -1.65 [-1.98 to -1.32] | -1.73 [-2.06 to -1.40]
  Week 12: number analyzed (Participants) | 34 | 31 | 45 | 44 | 45
  Week 12 | -1.38 [-1.78 to -0.97] | -1.67 [-2.08 to -1.26] | -1.94 [-2.29 to -1.59] | -2.00 [-2.36 to -1.65] | -2.12 [-2.47 to -1.77]

16. Secondary Outcome: Change From Baseline in DAS28-3 (CRP) at 4, 8 and 12 Weeks
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-3 (CRP) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed and hs-CRP. DAS28-3 (CRP) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 ln(CRP [mg/L] +1)*1.10+ 1.15. Total score range: 0-9.4. Higher score indicated more disease activity. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 47 | 47
  Week 4 | -0.61 [-0.90 to -0.32] | -0.93 [-1.22 to -0.64] | -1.09 [-1.35 to -0.84] | -1.01 [-1.27 to -0.76] | -0.88 [-1.14 to -0.62]
  Week 8: number analyzed (Participants) | 34 | 35 | 46 | 41 | 45
  Week 8 | -0.97 [-1.32 to -0.61] | -1.24 [-1.60 to -0.89] | -1.46 [-1.76 to -1.15] | -1.52 [-1.83 to -1.20] | -1.52 [-1.83 to -1.21]
  Week 12: number analyzed (Participants) | 34 | 31 | 45 | 44 | 45
  Week 12 | -1.14 [-1.52 to -0.77] | -1.53 [-1.91 to -1.15] | -1.82 [-2.14 to -1.50] | -1.83 [-2.15 to -1.50] | -1.82 [-2.15 to -1.50]

17. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at 4, 8 and 12 Weeks
Description: ACR20 was calculated as a 20% improvement in TJC and SJC and 20% improvement in 3 of the 5 remaining ACR core set measures: PtGA and PhGA, pain, disability, and an acute phase reactant which for this study was CRP or ESR. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4 | 30.8 [16.3 to 45.3] | 35.9 [20.8 to 51.0] | 42.0 [28.3 to 55.7] | 40.0 [26.4 to 53.6] | 37.5 [23.8 to 51.2]
  Week 8 | 46.2 [30.5 to 61.8] | 51.3 [35.6 to 67.0] | 58.0 [44.3 to 71.7] | 52.0 [38.2 to 65.8] | 64.6 [51.1 to 78.1]
  Week 12 | 51.3 [35.6 to 67.0] | 48.7 [33.0 to 64.4] | 66.0 [52.9 to 79.1] | 62.0 [48.5 to 75.5] | 70.8 [58.0 to 83.7]

18. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at 4, 8 and 12 Weeks
Description: ACR50 was calculated as a 50% improvement in TJC and SJC and 50% improvement in 3 of the 5 remaining ACR core set measures: PtGA and PhGA, pain, disability, and an acute phase reactant which for this study was CRP or ESR. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4 | 2.6 [0.0 to 7.5] | 10.3 [0.7 to 19.8] | 6.0 [0.0 to 12.6] | 6.0 [0.0 to 12.6] | 8.3 [0.5 to 16.2]
  Week 8 | 12.8 [2.3 to 23.3] | 23.1 [9.9 to 36.3] | 14.0 [4.4 to 23.6] | 22.0 [10.5 to 33.5] | 35.4 [21.9 to 48.9]
  Week 12 | 20.5 [7.8 to 33.2] | 25.6 [11.9 to 39.3] | 22.0 [10.5 to 33.5] | 40.0 [26.4 to 53.6] | 43.8 [29.7 to 57.8]

19. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at 4, 8 and 12 Weeks
Description: ACR70 was calculated as a 70% improvement in TJC and SJC and 70% improvement in 3 of the 5 remaining ACR core set measures: PtGA and PhGA, pain, disability, and an acute phase reactant which for this study was CRP or ESR. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
percentage of participants
  Week 4 | 0.0 [0.0 to 0.0] | 5.1 [0.0 to 12.1] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 4.2 [0.0 to 9.8]
  Week 8 | 2.6 [0.0 to 7.5] | 10.3 [0.7 to 19.8] | 0.0 [0.0 to 0.0] | 10.0 [1.7 to 18.3] | 6.3 [0.0 to 13.1]
  Week 12 | 5.1 [0.0 to 12.1] | 7.7 [0.0 to 16.1] | 6.0 [0.0 to 12.6] | 14.0 [4.4 to 23.6] | 10.4 [1.8 to 19.1]

20. Secondary Outcome: Change From Baseline in the Tender/Painful and Swollen Joint Counts at 4, 8 and 12 Weeks
Description: The TJC (28) included the following joints: shoulders, elbows, wrists, metatarsophalangeal (MCP) joints, PIP joints, and knees. This count was calculated from the TJC (68) assessed. The SJC (28) included the same joints as TJC (28), and was calculated from the SJC 66 assessed for swelling.Sixty eight (68) joints were assessed by a blinded joint assessor to determine the number of joints that were considered tender or painful. The 68 joints assessed were: temporomandibular, sternoclavicular, acromioclavicular; shoulder, elbow, wrist, MCPs, thumb interphalangeal, proximal interphalangeals, and distal interphalangeals; hip, knee, ankle, tarsus, metatarsophalangeals, great toe interphalangeal, proximal and distal interphalangeals combined. Sixty-six (66) joints were assessed for swelling, the same as those listed for TJC, excluding the right and left hip joints. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
joints
  SJC (28) at Week 4: number analyzed (Participants) | 37 | 38 | 49 | 49 | 47
  SJC (28) at Week 4 | -4.4 (6.01) | -4.8 (3.64) | -4.4 (3.76) | -5.0 (4.87) | -3.8 (4.25)
  SJC (28) at Week 8: number analyzed (Participants) | 35 | 35 | 46 | 46 | 47
  SJC (28) at Week 8 | -6.1 (6.75) | -6.0 (4.70) | -6.1 (4.80) | -7.0 (5.31) | -6.8 (5.75)
  SJC (28) at Week 12: number analyzed (Participants) | 34 | 31 | 45 | 45 | 45
  SJC (28) at Week 12 | -6.3 (5.61) | -6.8 (5.21) | -6.6 (5.38) | -8.1 (5.73) | -8.2 (6.01)
  TJC (28) at Week 4: number analyzed (Participants) | 37 | 38 | 49 | 49 | 47
  TJC (28) at Week 4 | -4.0 (5.99) | -4.9 (5.01) | -5.5 (5.12) | -4.8 (6.14) | -4.4 (5.36)
  TJC (28) at Week 8: number analyzed (Participants) | 35 | 35 | 46 | 46 | 47
  TJC (28) at Week 8 | -5.9 (7.16) | -6.9 (6.18) | -7.0 (5.83) | -7.5 (7.13) | -7.8 (6.72)
  TJC (28) at Week 12: number analyzed (Participants) | 34 | 31 | 45 | 45 | 45
  TJC (28) at Week 12 | -7.5 (6.39) | -8.6 (6.36) | -9.5 (6.14) | -9.9 (7.24) | -9.6 (6.65)
  SJC (66) at Week 4: number analyzed (Participants) | 37 | 38 | 49 | 49 | 47
  SJC (66) at Week 4 | -6.2 (10.82) | -6.5 (5.07) | -6.3 (5.27) | -8.6 (9.00) | -6.2 (8.00)
  SJC (66) at Week 8: number analyzed (Participants) | 35 | 35 | 46 | 46 | 47
  SJC (66) at Week 8 | -9.0 (10.87) | -8.2 (7.03) | -8.5 (6.74) | -11.0 (8.81) | -10.0 (9.92)
  SJC (66) at Week 12: number analyzed (Participants) | 34 | 31 | 45 | 45 | 45
  SJC (66) at Week 12 | -9.4 (9.92) | -9.6 (7.76) | -8.8 (7.11) | -12.5 (9.00) | -11.6 (10.19)
  TJC (68) at Week 4: number analyzed (Participants) | 37 | 38 | 49 | 49 | 47
  TJC (68) at Week 4 | -4.9 (11.28) | -8.7 (8.96) | -9.1 (8.45) | -9.1 (12.22) | -7.8 (9.60)
  TJC (68) at Week 8: number analyzed (Participants) | 35 | 35 | 46 | 46 | 47
  TJC (68) at Week 8 | -10.0 (13.41) | -10.9 (10.48) | -11.3 (9.46) | -14.0 (14.61) | -12.2 (11.40)
  TJC (68) at Week 12: number analyzed (Participants) | 34 | 31 | 45 | 45 | 45
  TJC (68) at Week 12 | -11.5 (12.24) | -13.5 (11.44) | -15.5 (11.30) | -18.1 (15.00) | -14.8 (11.98)

21. Secondary Outcome: Change From Baseline in High-Sensitivity C-Reactive Protein (Hs-CRP) at 4, 8 and 12 Weeks
Description: Serum samples were analyzed to determine the level of hs-CRP, which was an acute-phase reactant. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
mg/dL
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 47 | 47
  Week 4 | 0.22 [-0.17 to 0.60] | -0.15 [-0.53 to 0.23] | -0.66 [-1.00 to -0.32] | -0.66 [-1.00 to -0.32] | -0.65 [-1.00 to -0.31]
  Week 8: number analyzed (Participants) | 34 | 35 | 46 | 41 | 45
  Week 8 | 0.12 [-0.35 to 0.59] | 0.07 [-0.39 to 0.53] | -0.91 [-1.31 to -0.50] | -0.62 [-1.04 to -0.20] | -0.61 [-1.02 to -0.20]
  Week 12: number analyzed (Participants) | 34 | 31 | 46 | 44 | 45
  Week 12 | -0.07 [-0.54 to 0.39] | -0.23 [-0.71 to 0.25] | -0.74 [-1.14 to -0.34] | -0.68 [-1.09 to -0.27] | -0.64 [-1.04 to -0.23]

22. Secondary Outcome: Change From Baseline in the Physician's Global Assessment of Arthritis (PhGA) at 4, 8, and 12 Weeks
Description: The investigator assessed how the participant's overall arthritis appeared at the time of the visit. This was an evaluation based on the participant's disease symptoms, functional capacity and physical examination, and was independent of the participant's reported assessments of PtGA (patient's global assessment of arthritis). The investigator's response was recorded using a 100 mm visual analog scale (VAS), with the 0 mm end labeled "None" and the 100 mm end labeled "Extreme". Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  Week 4: number analyzed (Participants) | 37 | 37 | 49 | 49 | 47
  Week 4 | -14.30 [-20.06 to -8.54] | -18.54 [-24.31 to -12.78] | -22.51 [-27.53 to -17.49] | -18.34 [-23.34 to -13.33] | -18.06 [-23.20 to -12.92]
  Week 8: number analyzed (Participants) | 35 | 34 | 46 | 46 | 47
  Week 8 | -25.86 [-32.11 to -19.62] | -26.80 [-33.12 to -20.48] | -27.76 [-33.21 to -22.31] | -27.86 [-33.31 to -22.42] | -29.97 [-35.42 to -24.52]
  Week 12: number analyzed (Participants) | 34 | 30 | 46 | 45 | 45
  Week 12 | -28.16 [-34.59 to -21.74] | -30.28 [-36.98 to -23.58] | -33.05 [-38.61 to -27.49] | -34.27 [-39.86 to -28.68] | -36.34 [-41.95 to -30.73]

23. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Treatment-Related TEAEs
Description: AE was defined as any untoward medical occurrence in a clinical investigation participant administered a product or medical device, regardless of the causal relationship to study treatment. Treatment-emergent AEs (TEAEs) were defined as AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. Serious AEs (SAEs) were defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). AEs included SAEs and non-serious AEs. Causality to study treatment was determined by the investigator.
Time Frame: Baseline up to 28 calendar days after the last administration of the investigational product (about 21 months)
Population: The safety analysis population included the participants who received at least 1 dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofa 10 mg | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 43 | 39 | 50 | 50 | 48
Participants
  TEAEs (all causality) | 17 | 17 | 20 | 27 | 19 | 23
  TEAEs (treatment-related) | 8 | 6 | 12 | 8 | 8 | 6
  SAEs (all causality) | 1 | 1 | 1 | 1 | 1 | 3
  SAEs (treatment-related) | 0 | 0 | 1 | 0 | 0 | 0

24. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory evaluation included hematology, clinical chemistry, and urinalysis. Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell, platelet and white blood cell count, neutrophils, eosinophils, monocytes, basophils and lymphocytes), chemistry (blood urea nitrogen, creatinine, sodium, potassium, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein and serum pregnancy test [for all female participants]) and urine (urine pregnancy test [for all female participants]). Each parameter was evaluated against commonly used and widely accepted criteria. Clinical significance of laboratory parameters was determined at the investigator's discretion. The investigator judged the abnormality.
Time Frame: Baseline up to 28 calendar days after the last administration of the investigational product (about 21 months)
Population: The safety analysis population included all participants who received at least 1 dose of investigational drug and were evaluable for laboratory abnormalities.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofa 10 mg | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 38 | 43 | 39 | 50 | 49 | 48
Participants | 30 | 32 | 30 | 36 | 41 | 38

25. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-sepcified Criteria
Description: Vital Signs tests included sitting systolic blood pressure (SBP) and diastolic blood pressure (DBP) and pulse rate. Vital signs categorical summarization criteria were 1), systolic BP (SBP) <90 millimeters of mercury (mm Hg) or change from baseline (Chg) >=30mm Hg; diastolic BP (DBP) <50mm Hg or change from baseline >=20mm Hg; 2), pulse rate <40bpm or > 120bpm.
Time Frame: Baseline up to 28 calendar days after the last administration of the investigational product (about 21 months)
Population: The safety analysis population included all participants who received at least 1 dose of investigational drug and had evaluable vital signs data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofa 10 mg | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 38 | 43 | 39 | 50 | 49 | 48
Participants
  Sitting Diastolic BP < 50 mm Hg | 1 | 0 | 0 | 0 | 0 | 0
  Sitting Pulse Rate < 40 bpm | 0 | 0 | 0 | 0 | 0 | 0
  Sitting Pulse Rate > 120 bpm | 0 | 0 | 0 | 0 | 0 | 0
  Sitting Systolic BP < 90 mm Hg | 0 | 0 | 0 | 0 | 0 | 0
  Increase: Sitting Systolic BP Chg>= 30 mm Hg | 0 | 0 | 1 | 1 | 0 | 1
  Increase: Sitting Diastolic BP Chg >= 20 mmHg | 1 | 2 | 3 | 0 | 1 | 2
  Decrease: Sitting Systolic BP Chg >= 30 mm Hg | 2 | 3 | 0 | 2 | 3 | 3
  Decrease: Sitting Diastolic BP Chg >= 20 mm Hg | 2 | 4 | 2 | 4 | 3 | 2

26. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-sepcified Criteria
Description: ECG evaluation included: PR interval, time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS interval), time between the start of the Q wave and the end of the T wave in the heart's electrical cycle (QT interval), QT interval corrected for heart rate using Fridericia's formula (QTcF interval), and QTc calculated using Bazett's correction factor (QTcB interval).
Time Frame: Baseline up to 28 calendar days after the last administration of the investigational product (about 21 months)
Population: The safety analysis population included all participants who received at least 1 dose of investigational drug and had evaluable ECG data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofa 10 mg | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 38 | 43 | 39 | 50 | 49 | 48
Participants
  PR interval >=300 msec | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration >=140 msec | 0 | 0 | 0 | 0 | 0 | 0
  QT interval >=500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcB interval >=450 and <480 msec | 5 | 4 | 5 | 4 | 5 | 13
  QTcB interval >=480 and <500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcB interval >=500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval >=450 and <480 msec | 0 | 1 | 1 | 0 | 1 | 4
  QTcF interval >=480 and <500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval >=500 msec | 0 | 0 | 0 | 0 | 0 | 0
  PR interval increase>=25/50% | 0 | 0 | 0 | 0 | 1 | 0
  QRS duration increase>=50% | 0 | 0 | 0 | 0 | 0 | 0
  QTcB interval increase>=30 and increase <60 msec | 3 | 6 | 9 | 3 | 4 | 7
  QTcB interval increase>=60 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval increase>=30 and increase <60 msec | 2 | 4 | 5 | 0 | 5 | 5
  QTcF interval increase>=60 msec | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Urinalysis Data Meeting Pre-specified Criteria
Description: The urine sample was collected for central laboratory urinalysis and urine microscopy. The urinalysis included pH, protein, glucose, erythrocytes, leukocytes, ketones, nitrite, urobilinogen, urine bilirubin, urine hemoglobin, leukocyte esterase, granular casts, hyaline casts, bacteria, atypical, needle-like crystals urine, specific gravity, microscopy and urine albumin test.
Time Frame: Baseline up to 28 calendar days after the last administration of the investigational product (about 21 months)
Population: The safety analysis population included all participants who received at least 1 dose of investigational drug and had evaluable urinalysis data
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofa 10 mg | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 38 | 43 | 39 | 50 | 49 | 48
Participants
  Specific gravity <1.003 | 0 | 0 | 0 | 0 | 0 | 0
  Specific gravity >1.030 | 3 | 0 | 0 | 3 | 2 | 2
  pH <4.5 | 0 | 0 | 0 | 0 | 0 | 0
  pH >8 | 0 | 0 | 0 | 0 | 0 | 0
  Urine glucose >=1 | 0 | 0 | 4 | 2 | 2 | 2
  Ketones >=1 | 3 | 0 | 1 | 2 | 1 | 1
  Urine protein >=1 | 0 | 0 | 0 | 0 | 1 | 0
  Urine hemoglobin >=1 | 7 | 5 | 6 | 5 | 12 | 6
  Urobilinogen >=1 | 1 | 0 | 0 | 0 | 0 | 1
  Urine bilirubin >=1 | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite >=1 | 3 | 5 | 3 | 1 | 9 | 11
  Leukocyte esterase >=1 | 16 | 15 | 14 | 14 | 19 | 19
  Urine erythrocytes(/HPF) >=20: number analyzed (Participants) | 32 | 32 | 32 | 34 | 37 | 35
  Urine erythrocytes(/HPF) >=20 | 1 | 2 | 3 | 1 | 3 | 3
  Urine leukocytes (/HPF) >=20: number analyzed (Participants) | 30 | 42 | 38 | 47 | 48 | 43
  Urine leukocytes (/HPF) >=20 | 4 | 3 | 2 | 2 | 7 | 7
  Granular casts (/LPF) >1: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 0
  Granular casts (/LPF) >1 | 1 | 1 | 0 | 0 | 0 | 0
  Hyaline Casts (/LPF): number analyzed (Participants) | 7 | 11 | 10 | 16 | 9 | 8
  Hyaline Casts (/LPF) | 4 | 4 | 6 | 7 | 4 | 3
  Bacteria >20: number analyzed (Participants) | 23 | 29 | 22 | 34 | 31 | 33
  Bacteria >20 | 0 | 0 | 0 | 0 | 0 | 0
  Atypical, needle-like crystals urine >=1 | 0 | 0 | 0 | 0 | 2 | 0

28. Secondary Outcome: Change From Baseline in the Patient's Assessment of Arthritis Pain (PAAP) Visual Analogue Scale (VAS) at Weeks 4, 8, 12
Description: Patients assess the severity of their arthritis pain using a 100 mm VAS by placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponds to the magnitude of their pain. This assessment was performed early in the clinic visit and before the participant had extensive contact with site personnel and/or Investigator. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 49 | 47
  Week 4 | -12.8 (18.85) | -11.5 (19.44) | -16.8 (20.19) | -9.5 (16.10) | -11.3 (21.22)
  Week 8: number analyzed (Participants) | 35 | 35 | 46 | 46 | 47
  Week 8 | -22.4 (20.05) | -15.4 (21.32) | -22.2 (18.88) | -20.5 (23.70) | -23.5 (20.42)
  Week 12: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  Week 12 | -25.9 (26.39) | -21.4 (25.03) | -23.0 (21.46) | -25.7 (24.02) | -31.08 (23.70)

29. Secondary Outcome: Change From Baseline in the Patient Global Assessment of Arthritis (PtGA) VAS at Weeks 4, 8, 12
Description: Patients answer the following question: "Considering all the ways your arthritis affects you, how are you feeling today?" The patient's response is recorded using a 100 mm VAS. This assessment was performed early in the clinic visit and before the participant had extensive contact with site personnel and/or Investigator. The higher score indicated more severe disease. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  Week 4: number analyzed (Participants) | 37 | 38 | 50 | 50 | 47
  Week 4 | -12.0 (21.55) | -10.0 (16.68) | -14.9 (20.52) | -10.7 (19.11) | -13.7 (20.29)
  Week 8: number analyzed (Participants) | 35 | 35 | 46 | 46 | 47
  Week 8 | -24.9 (21.25) | -13.1 (23.47) | -19.6 (19.60) | -22.2 (27.34) | -25.3 (20.74)
  Week 12: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  Week 12 | -25.9 (25.03) | -20.0 (23.12) | -19.7 (25.71) | -26.5 (25.23) | -34.2 (22.81)

30. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire - Disability Index (HAQ-DI) at Weeks 4, 8, and 12
Description: The HAQ-DI was defined as participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: The analysis population included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (PF-06650833, tofacitinib, or placebo).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  Week 4: number analyzed (Participants) | 37 | 38 | 49 | 49 | 47
  Week 4 | -0.2 (0.46) | -0.2 (0.44) | -0.3 (0.40) | -0.2 (0.43) | -0.3 (0.49)
  Week 8: number analyzed (Participants) | 35 | 35 | 46 | 46 | 47
  Week 8 | -0.4 (0.47) | -0.4 (0.54) | -0.4 (0.41) | -0.4 (0.56) | -0.5 (0.59)
  Week 12: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  Week 12 | -0.5 (0.47) | -0.5 (0.60) | -0.5 (0.48) | -0.5 (0.66) | -0.6 (0.59)

31. Secondary Outcome: Change From Baseline in the 36 Item Short Form Health Survey (SF-36) Version 2 (Acute) 8 Domain Scores at Week 12
Description: The SF-36 version 2 (acute) is a 36 item generic health status measure. It measures 8 general health domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The SF-36 summary scores range from 0-100, with higher scores representing better self-reported health. This was performed early in the clinic visit and before the participant had extensive contact with site personnel and/or Investigator. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  Physical functioning domain: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  Physical functioning domain | 3.311 (11.5441) | 4.885 (8.4161) | 6.318 (8.6700) | 5.412 (9.7871) | 7.322 (11.2219)
  Role-physical domain: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  Role-physical domain | 6.316 (9.7393) | 5.773 (10.0629) | 6.173 (8.5158) | 6.151 (9.8448) | 6.734 (9.3707)
  Bodily pain domain: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  Bodily pain domain | 7.840 (7.2950) | 6.543 (9.3835) | 7.280 (8.1633) | 7.071 (9.6901) | 10.422 (8.6959)
  General health domain: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  General health domain | 5.775 (6.7414) | 5.531 (6.4448) | 4.856 (6.5230) | 4.916 (8.4424) | 7.046 (8.7992)
  Vitality domain: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  Vitality domain | 8.717 (8.0179) | 7.049 (9.9149) | 7.354 (9.9326) | 6.453 (10.2902) | 8.182 (8.7136)
  Social function domain: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  Social function domain | 5.061 (11.6125) | 6.418 (11.6517) | 6.430 (12.2952) | 6.095 (12.1659) | 8.485 (9.2070)
  Role-emotional domain: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  Role-emotional domain | 7.683 (11.2028) | 4.396 (11.1492) | 5.103 (12.5489) | 6.730 (12.7335) | 6.646 (11.4190)
  Mental health domain: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  Mental health domain | 7.497 (11.8826) | 5.161 (11.7376) | 5.661 (13.7839) | 7.080 (12.9887) | 8.866 (10.4266)

32. Secondary Outcome: Change From Baseline in the Physical Component Score (PCS) and Mental Component Score (MCS) at Week 12
Description: The SF 36 version 2 (acute) is a 36 item generic health status measure. It measures 8 general health domains. These domains can also be summarized as physical component score (PCS) and mental component score (MCS). The PCS and MCS summary scores range from 0-100, with higher scores representing better self-reported health. The lower the score the more disability. This was performed early in the clinic visit and before the participant had extensive contact with site personnel and/or Investigator. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  PCS: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  PCS | 4.635 (7.8031) | 5.728 (7.4254) | 6.304 (7.6091) | 5.212 (8.0162) | 7.476 (8.3473)
  MCS: number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
  MCS | 7.995 (11.5950) | 5.241 (10.4860) | 5.425 (13.6873) | 6.749 (12.0657) | 7.759 (9.4263)

33. Secondary Outcome: Change From Baseline in the European Quality of Life 5 Dimensions-3 Level (EQ-5D-3L) Score at Week 12
Description: The EQ-5D-3L health state profile is a patient completed questionnaire designed to assess impact on health related quality of life in 5 domains: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Additionally, scores from the 5 domains might have been used to calculate a single index value, also known as a utility score. The validity and reliability of the EQ-5D-3L have been established in a number of disease states, including RA. EQ-5D-3L scores marked health status from 0 and 100. There were notes at the both ends of the scale that the bottom rate (0) corresponded to " the worst health you could imagine", and the highest rate (100) corresponded to "the best health you could imagine". Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 39 | 39 | 50 | 50 | 48
units on a scale
  EQ visual analogue scale (VAS) score: number analyzed (Participants) | 34 | 31 | 46 | 44 | 45
  EQ visual analogue scale (VAS) score | 13.265 (18.8540) | 11.129 (24.6181) | 11.913 (20.3795) | 20.909 (24.5895) | 20.778 (20.6792)
  Index value: number analyzed (Participants) | 34 | 31 | 45 | 45 | 45
  Index value | 0.132 (0.2030) | 0.056 (0.1957) | 0.118 (0.1661) | 0.143 (0.2445) | 0.190 (0.2201)

34. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Total Score at Week 12
Description: The FACIT-F is a patient completed questionnaire consisting of 13 items that assess fatigue. Instrument scoring yields a range from 0 to 52, with higher scores representing better patient status (less fatigue). This questionnaire was performed early in the clinic visit and before the participant had extensive contact with site personnel and/or investigator. Tofacitinib was included in this study as an active control. The efficacy endpoint for the tofatinicib arm was an exploratory endpoint and neither primary nor secondary endpoints.
Time Frame: Baseline and Week 12
Population: The analysis population included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (PF-06650833, tofacitinib, or placebo). It was pre-specified in the protocol to not summarize this efficacy endpoint for Tofa arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
Number analyzed (Participants) | 34 | 31 | 46 | 45 | 45
units on a scale | 8.4 (8.76) | 4.6 (10.92) | 6.8 (8.33) | 7.2 (11.45) | 9.5 (9.68)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 calendar days after the last administration of the investigational product (about 21 months)
Description: The same event may appear as both an AE and a SAE. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Placebo | Tofa 10 mg | PF-06650833 20 mg | PF-06650833 60 mg | PF-06650833 200 mg | PF-06650833 400 mg
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/43 | 0/39 | 0/50 | 0/50 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/39 | 1/43 | 1/39 | 1/50 | 1/50 | 3/48
Other Adverse Events (participants affected / at risk) | 10/39 | 8/43 | 12/39 | 11/50 | 9/50 | 11/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=39) | Tofa 10 mg (N=43) | PF-06650833 20 mg (N=39) | PF-06650833 60 mg (N=50) | PF-06650833 200 mg (N=50) | PF-06650833 400 mg (N=48)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0/48 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=39) | Tofa 10 mg (N=43) | PF-06650833 20 mg (N=39) | PF-06650833 60 mg (N=50) | PF-06650833 200 mg (N=50) | PF-06650833 400 mg (N=48)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2 | 0 | 2 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 2 | 1 | 3
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 4 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3 | 4 | 2 | 1 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 1 | 2 | 1
Headache (Nervous system disorders) | 2 | 0 | 1 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT02996500/SAP_000.pdf
  • Study Protocol (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT02996500/Prot_001.pdf